CLINICAL TRIAL: NCT02749890
Title: A Randomized, Active-controlled, Open Label, 2-treatment Arm, and Multicenter Study Comparing the Efficacy and Safety of Insulin Glargine/Lixisenatide Combination to Lixisenatide on Top of OADs in Japanese Patients With Type 2 DM With an Extension Period
Brief Title: Efficacy and Safety of the Insulin Glargine/Lixisenatide Fixed Ratio Combination (LixiLan) to Lixisenatide on Top of Oral Anti-diabetic Drugs (OADs) With Type 2 Diabetes in Japan
Acronym: LIXILAN JP-O1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC14112; U1111-1176-8357 (Other: UTN)
Record Dates: First submitted 2016-04-20; First posted 2016-04-25 (Estimated); Last update posted 2020-06-16 (Actual); Status verified 2018-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; lixisenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LixiLan (Experimental): LixiLan (insulin glargine/lixisenatide fixed ratio combination) is injected subcutaneously (under the skin) once daily. Dose is individually adjusted.
  Background therapy with OADs (except dipeptidyl-peptidase-4 inhibitor) should be continued during the treatment period.
  Interventions: Drug: Insulin glargine/Lixisenatide (HOE901/AVE0010); Drug: Oral anti-diabetic drugs
- lixisenatide (Active Comparator): Lixisenatide (AVE0010) is injected subcutaneously (under the skin) once daily. It will be initiated with Dose 1 for 1 week and then continue with Dose 2 for 1 week followed by the maintenance dose of Dose 3 up to the end of treatment period.
  Background therapy with OADs (except dipeptidyl-peptidase-4 inhibitor) should be continued during the treatment period.
  Interventions: Drug: Lixisenatide (AVE0010); Drug: Oral anti-diabetic drugs

INTERVENTIONS:
Drug: Insulin glargine/Lixisenatide (HOE901/AVE0010) — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Other Names: LixiLan
  Arms: LixiLan
Drug: Lixisenatide (AVE0010) — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Arms: lixisenatide
Drug: Oral anti-diabetic drugs — Pharmaceutical form: tablet
  Route of administration: Oral

SUMMARY:
Primary Objective:

To compare LixiLan to lixisenatide in glycated hemoglobin (HbA1c) change from baseline to Week 26 in patients with type 2 diabetes mellitus.

Secondary Objective:

To compare the overall efficacy and safety of LixiLan to lixisenatide (with or without OADs) over a 52 week treatment period in patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Approximately 55 weeks: an up-to 2-week screening period, a 26-week randomized open-label treatment period, a 26-week safety extension treatment period and a 3-day post-treatment safety follow up period.

ELIGIBILITY:
Inclusion criteria :

* Patient with type 2 diabetes mellitus (T2DM) diagnosed for at least 1 year before the screening visit, receiving 1 or 2 OADs that can be biguanide, thiazolidinedione, alpha-glucosidase-inhibitor, sodium glucose co-transporter 2 inhibitor; sulfonylurea, rapid-acting insulin secretagogue, or dipeptidyl-peptidase-4 inhibitor.
* Signed written informed consent.

Exclusion criteria:

* At the screening visit: age <20 years.
* At the screening visit: HbA1c <7.5% or >10%.
* At the screening visit: fasting plasma glucose (FPG) >250 mg/dL (13.8 mmol/L).
* Pregnancy or lactation, women of childbearing potential with no effective contraceptive method.
* Use of oral or injectable glucose-lowering agents other than those stated in the inclusion criteria during the 3 months before the screening visit.
* Previous treatment with insulin (except for short-term treatment due to intercurrent illness including gestational diabetes at the discretion of the trial physician).
* Laboratory findings at the screening visit, including:
* Amylase and/or lipase >3 times the upper limit of the normal laboratory range (ULN),
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 ULN,
* Calcitonin ≥20 pg/mL (5.9 pmol/L),
* Positive serum pregnancy test.
* Contraindication to use of lixisenatide according to the local labeling. History of hypersensitivity to any glucagon-like peptide-1 receptor agonist (GLP-1RA) or to metacresol.
* Contraindication to use of insulin glargine according to the local labeling. History of hypersensitivity to insulin glargine or to any of the excipients.
* Patient who has a severe renal function impairment with estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m^2 or end-stage renal disease for patient not treated with metformin.
* Personal or immediate family history of medullary thyroid cancer (MTC) or genetic condition that predisposes to MTC (eg, multiple endocrine neoplasia syndromes).
* History of pancreatitis (unless pancreatitis was related to gallstones and cholecystectomy has been performed), pancreatitis during previous treatment with incretin therapies, chronic pancreatitis, pancreatectomy, stomach/gastric surgery.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2016-05-09 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c | Baseline, 26 weeks

SECONDARY OUTCOMES:
Percentage of patients reaching HbA1c <7% or ≤6.5% | 26 weeks
Change from baseline in fasting plasma glucose | Baseline, 26 weeks
Change in from baseline in 7 point self-monitored plasma profiles | Baseline, 26 weeks
Percentage of patients reaching HbA1c <7% with no body weight gain | 26 weeks
Change from baseline in body weight | Baseline, 26 weeks
Percentage of patients requiring a rescue therapy | 26 weeks
Change in daily dose of insulin glargine for the combination group | Day 1, 26 weeks
Number of hypoglycemic events | 26 weeks, 52 weeks
Number of adverse events | 26 weeks, 52 weeks
Measurement of anti-lixisenatide antibodies from baseline | Baseline, 26 weeks, 52 weeks
Measurement of anti-insulin antibodies from baseline | Baseline, 26 weeks, 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (61):
- Japan (61):
  - Investigational Site Number 392002, Adachi-Ku
  - Investigational Site Number 392009, Arakawa-Ku
  - Investigational Site Number 392025, Atsugi-Shi
  - Investigational Site Number 392060, Bunkyō City
  - Investigational Site Number 392024, Chiba
  - Investigational Site Number 392011, Chigasaki-Shi
  - Investigational Site Number 392013, Chiyoda-Ku
  - Investigational Site Number 392052, Chiyoda-Ku
  - Investigational Site Number 392003, Chūōku
  - Investigational Site Number 392017, Chūōku
  - Investigational Site Number 392008, Fujimi-Shi
  - Investigational Site Number 392054, Fukuoka
  - Investigational Site Number 392094, Fukuoka
  - Investigational Site Number 392059, Hachioji-Shi
  - Investigational Site Number 392083, Hakodate-Shi
  - Investigational Site Number 392048, Hamamatsu
  - Investigational Site Number 392079, Hiki-Gun
  - Investigational Site Number 392057, Iruma-Shi
  - Investigational Site Number 392022, Ise-Shi
  - Investigational Site Number 392023, Isehara-Shi
  - Investigational Site Number 392020, Izumisano
  - Investigational Site Number 392066, Kashiwa-Shi
  - Investigational Site Number 392006, Kasugai-Shi
  - Investigational Site Number 392053, Kawagoe-Shi
  - Investigational Site Number 392065, Kawagoe-Shi
  - Investigational Site Number 392007, Kawaguchi-Shi
  - Investigational Site Number 392062, Kawaguchi-Shi
  - Investigational Site Number 392077, Kawasaki-Shi
  - Investigational Site Number 392082, Kawasaki-Shi
  - Investigational Site Number 392031, Kitakyushu-Shi
  - Investigational Site Number 392041, Kitakyusyu-Shi
  - Investigational Site Number 392068, Kitakyusyu-Shi
  - Investigational Site Number 392044, Koga-Shi
  - Investigational Site Number 392001, Koriyama-Shi
  - Investigational Site Number 392032, Kurume-Shi
  - Investigational Site Number 392088, Maebashi
  - Investigational Site Number 392014, Mitaka-Shi
  - Investigational Site Number 392042, Mito
  - Investigational Site Number 392078, Mito
  - Investigational Site Number 392026, Nagoya
  - Investigational Site Number 392080, Okayama
  - Investigational Site Number 392040, Oyama-Shi
  - Investigational Site Number 392038, Sagamihara-Shi
  - Investigational Site Number 392069, Saijo-Shi
  - Investigational Site Number 392030, Saitama-Shi
  - Investigational Site Number 392047, Sapporo
  - Investigational Site Number 392015, Satsumasendai-Shi
  - Investigational Site Number 392004, Sendai
  - Investigational Site Number 392034, Shimotsuke-Shi
  - Investigational Site Number 392037, Shizuoka
  - Investigational Site Number 392081, Shizuoka
  - Investigational Site Number 392019, Shobara-Shi
  - Investigational Site Number 392018, Shunan-Shi
  - Investigational Site Number 392027, Suita-Shi
  - Investigational Site Number 392056, Taito-Ku
  - Investigational Site Number 392051, Takatsuki-Shi
  - Investigational Site Number 392061, Tokorozawa-Shi
  - Investigational Site Number 392029, Toyonaka-Shi
  - Investigational Site Number 392093, Ube-Shi
  - Investigational Site Number 392067, Yatsushiro-Shi
  - Investigational Site Number 392035, Zentsuji-Shi

REFERENCES:
- [Result] Watada H, Takami A, Spranger R, Amano A, Hashimoto Y, Niemoeller E. Efficacy and Safety of 1:1 Fixed-Ratio Combination of Insulin Glargine and Lixisenatide Versus Lixisenatide in Japanese Patients With Type 2 Diabetes Inadequately Controlled on Oral Antidiabetic Drugs: The LixiLan JP-O1 Randomized Clinical Trial. Diabetes Care. 2020 Jun;43(6):1249-1257. doi: 10.2337/dc19-2452. Epub 2020 Apr 15. PMID 32295808